CLINICAL TRIAL: NCT05449119
Title: Loss of Autonomy in the Elderly: Relationships Between Gut Microbiota Diversity, Nutrition and Cognitive and Sensory-motor Disturbances in "Small Eaters" and "Non Small Eaters"
Acronym: ALMICO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DALLE CHU 2020
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Elderly Small Eater
MeSH Terms: interventions — Defecation; Blood Specimen Collection; Body Mass Index; Food; Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non small eaters: Elderly subjects who are not malnourished
  Interventions: Biological: Fecal and blood sampling and collection of nutritional, cognitive and sensorimotor data; Other: Body Mass Index (BMI); Other: 24-hour food and beverage record; Other: Mini Nutritional assessment (MNA); Other: Measurement of muscle mass by bioelectrical impedance analysis (except for participants with a pacemaker); Other: Measurement of sensorimotor functions; Other: Measurement of cognitive functions
- Small eaters: Elderly subjects with loss of appetite
  Interventions: Biological: Fecal and blood sampling and collection of nutritional, cognitive and sensorimotor data; Other: Body Mass Index (BMI); Other: 24-hour food and beverage record; Other: Mini Nutritional assessment (MNA); Other: Measurement of muscle mass by bioelectrical impedance analysis (except for participants with a pacemaker); Other: Measurement of sensorimotor functions; Other: Measurement of cognitive functions

INTERVENTIONS:
Biological: Fecal and blood sampling and collection of nutritional, cognitive and sensorimotor data — at T0, T3 months, T6 months, T9 months and T12 months
Other: Body Mass Index (BMI) — Calculation of BMI with height measurement by heel-knee distance measurement at T0, T3 months, T6 months, T9 months and T12 months
Other: 24-hour food and beverage record — at T0, T3 months, T6 months, T9 months and T12 months
Other: Mini Nutritional assessment (MNA) — at T0, T3 months, T6 months, T9 months and T12 months
Other: Measurement of muscle mass by bioelectrical impedance analysis (except for participants with a pacemaker) — at T0, T3 months, T6 months, T9 months and T12 months
Other: Measurement of sensorimotor functions — at T0, T3 months, T6 months, T9 months and T12 months
Other: Measurement of cognitive functions — at T0, T3 months, T6 months, T9 months and T12 months

SUMMARY:
Older adults currently make up 25% of the population in France, and future health expenditures will be largely related to the consequences of aging. Normal aging is associated with a progressive decrease in cognitive and sensorimotor function, malnutrition and/or under-nutrition and intestinal dysbiosis (i.e. changes in the composition and/or stability of the microbiota). Furthermore, admission to long-term care facilities such as Etablissement d'Hébergement pour Personnes Agées Dépendantes (EHPAD) leads to drastic changes in lifestyle in terms of (i) nutrition and (ii) motor functions. These modifications can influence the composition of the intestinal microbiota and its temporal evolution.

We will study the relationship between the deterioration of cognitive and sensorimotor function, diet and intestinal well-being (i.e. microbiota) of a cohort of older adults (>75 years) defined as "small eaters" from their admission in EHPAD at the University Hospital of Dijon. This study will be carried out by a unique French multidisciplinary consortium that includes academics and health professionals, who will be able to specify the criteria defining the "small eaters" and to envisage suitable dietary strategies aiming to preserve their nutritional status and intestinal well-being. The final goal is to improve quality of life at home by prolonging autonomy and independence, and thus to deferring admission to an EHPAD for as long as possible.

The objective of this study is to build a cohort of elderly "small eaters" and a cohort of elderly "non small eaters". These patients will be followed over a period of one year. The evolution of the composition of the intestinal microbiota will be determined in order to establish the existing relations between the composition of digestive microbiota, the nutritional state, and cognitive and sensorimotor function.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent and has not objected to being included in the study, or if necessary, oral consent of an appointed legal representative.
* A person over 75 years of age residing in an EHPAD who may be under guardianship or curatorship.
* A person over 75 years of age with a loss of appetite (i.e. a small eater) residing in an EHPAD, who may be under guardianship or curatorship.

Exclusion Criteria:

* Person not affiliated to national health insurance
* Elderly person with an infectious syndrome at the time of admission;
* Elderly person with diarrhoea (infectious or not) at the time of admission;
* Elderly person receiving recently prescribed antimicrobials at the time of admission (antibiotics or antifungals)
* Elderly person with celiac disease and/or Crohn's disease.
* Person under a measure of limited judicial protection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people over 75 years old residing in EHPAD with a loss of appetite or not malnourished.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of the alpha diversity of the microbiota and the intestinal mycobiota | up to T12 months
  Measure indicating the diversity of a single sample
Measurement of the beta diversity of the microbiota and the intestinal mycobiota | up to T12 months
  Measure of species diversity between samples

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France